CLINICAL TRIAL: NCT02606513
Title: Opacification of the Upper Urinary Tract With MR Urography Compared to CT Urography
Brief Title: MR Urography vs CT Urography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Mazen Sudah, Senior Radiology Consultant, Kuopio University Hospital
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: MR_CT_URO
Record Dates: First submitted 2015-11-12; First posted 2015-11-17 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Neoplasms
Keywords: Computed Tomography Urography; Magnetic Resonance Urography
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Comparison of CTU vs MRU (Experimental): CTU is the primary test of choice for the evaluation of the UUT. The performance of MRU will be compared to that of CTU in the same patient population
  Interventions: Other: MR Urography; CT Urography

INTERVENTIONS:
Other: MR Urography; CT Urography

SUMMARY:
Tumors of the UUT are rare and usually presenting as micro- or macrohematuria either symptomatic or asymptomatic. Rapid advances in CT technology accelerated the research into the application of this new technology in the evaluation of the UUT and readily proved to be superior to other imaging modalities. Nevertheless the increase in radiation dose is a major issue of concern. Initial research into the utility of MRI in the evaluation of the UUT was promising, yet the success of CT together with the cost, limited availability and the longer duration of MR urography (MRU) examination, nearly halted the investigations into the feasibility of MRU which is unfortunate as MRU is a safe alternative to CT.

DETAILED DESCRIPTION:
Images from a MDCT scan are reconstructed into thin slices which can be viewed in any orientation with similar image quality compared to the original axial images. Completely isotropic resolution in 16- to 64-slice CT can be achieved using 0.5- to 0.625-mm slice thickness. Resulting images have high noise levels unless the tube load is increased considerably. In most clinical situations a near-isotropic resolution with 1.0- to 1.5-mm effective slice thickness suffices for high-quality images created in any plane using MPR.

‬Research into the accuracy of CTU in the evaluation of possible UUT malignancy soon proved CTU to be a very sensitive and specific method with pooled sensitivity of 96% (range 88-100%), and pooled specificity of 99% (range 93-100%). Furthermore direct comparison confirmed the superiority of CTU over IVU in terms of sensitivity and specificity.

In order to reduce confusion in terminology, the European Society of Urogenital Radiology's (ESUR) CTU Working Group proposes to define CTU as "a diagnostic examination optimized for imaging the kidneys, ureters and bladder. The examination involves the use of MDCT with thin-slice imaging, intravenous administration of a contrast medium, and imaging in the excretory phase." ESUR guideline comprehensively addresses all aspects of CTU based on extensive literature review and on the opinion of leading researchers in this field.‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬ To begin with, hydrating the patient is beneficial to reduce possible contrast induced nephropathy especially in otherwise dehydrated or not well hydrated patient, and at the same time provides negative bowel contrast medium. Usually 1 liter of water is slowly ingested during a period of 20-60 minutes before the CTU examination or alternatively a maximum of 500 ml slow intravenous drip-infusion of 0.9% saline may be used in patients who cannot tolerate per oral hydration. Nevertheless the ESUR guideline also concludes that the net benefit of intravenous saline bolus hydration is probably minimal and its routine use is thus not advocated. Bowel preparation with positive contrast will inevitably interfere with the interpretation especially in the demonstrative quality of reformatted images and is not recommended. In diuretic-enhanced CT urography, the patients are asked to empty their bladder before starting the CTU examination, nevertheless the ESUR guidelines have no stand on this issue. The use of compression pads is a routine practice in IVU and consequently it was thought that this maneuver can be transferred to the CTU protocol. However after evaluating of the available evidence ESUR guideline do not advocate the use of compression.

Patients are scanned in supine position. Prone position is not advocated to be used routinely but can be used in special cases e.g. to reduce layering effects of the contrast medium, especially when the renal collecting system is dilated.

After the introduction of the rapid MDCT technology it became clear that this new imaging modality is more accurate than IVU in the initial workout of a wide range of UUT pathology. Images from a MDCT scan are reconstructed into thin slices which can be viewed in any orientation with similar image quality compared to the original axial images. Completely isotropic resolution in 16- to 64-slice CT can be achieved using 0.5- to 0.625-mm slice thickness. Resulting images have high noise levels unless the tube load is increased considerably. In most clinical situations a near-isotropic resolution with 1.0- to 1.5-mm effective slice thickness suffices for high-quality images created in any plane using MPR.

‬Research into the accuracy of CTU in the evaluation of possible UUT malignancy soon proved CTU to be a very sensitive and specific method with pooled sensitivity of 96% (range 88-100%), and pooled specificity of 99% (range 93-100%). Furthermore direct comparison confirmed the superiority of CTU over IVU in terms of sensitivity and specificity.

In order to reduce confusion in terminology, the European Society of Urogenital Radiology's (ESUR) CTU Working Group proposes to define CTU as "a diagnostic examination optimized for imaging the kidneys, ureters and bladder. The examination involves the use of MDCT with thin-slice imaging, intravenous administration of a contrast medium, and imaging in the excretory phase.". ESUR guideline comprehensively addresses all aspects of CTU based on extensive literature review and on the opinion of leading researchers in this field.‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬ To begin with, hydrating the patient is beneficial to reduce possible contrast induced nephropathy especially in otherwise dehydrated or not well hydrated patient, and at the same time provides negative bowel contrast medium. Usually 1 liter of water is slowly ingested during a period of 20-60 minutes before the CTU examination or alternatively a maximum of 500 ml slow intravenous drip-infusion of 0.9% saline may be used in patients who cannot tolerate per oral hydration. Nevertheless the ESUR guideline also concludes that the net benefit of intravenous saline bolus hydration is probably minimal and its routine use is thus not advocated. Bowel preparation with positive contrast will inevitably interfere with the interpretation especially in the demonstrative quality of reformatted images and is not recommended. In diuretic-enhanced CT urography, the patients are asked to empty their bladder before starting the CTU examination, nevertheless the ESUR guidelines have no stand on this issue. The use of compression pads is a routine practice in IVU and consequently it was thought that this maneuver can be transferred to the CTU protocol. However after evaluating of the available evidence ESUR guideline do not advocate the use of compression.

‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬The first popular CTU protocol is the single-bolus 3-phase technique. After hydration, a low-dose unenhanced CT is acquired from the top of kidneys to the base of the bladder, followed first by low-dose diuretic and 1-2 minutes later by contrast injection. Imaging strategy after the administration of contrast material is controversial with different protocols available aimed mainly to detect or rule out possible malignancies and no scientific evidence is available on the superiority of specific protocols. Contrast enhanced abdominal scan can be obtained at corticomedullary phase (25-35 s delay after start of contrast injection) or at nephrographic (delay of 90-110 s) or with a combination of nephrographic-corticomedullary (so called dose-efficient or arterial-nephrographic-corticomedullary phase after splitting of the contrast injection into two or three bolus in modified protocols. The third excretory phase (240-480 s delay) is the most important scan with the purpose of achieving excellent endoluminal opacification, preferably with some UUT dilatation. Even better results are reported if acquisition is further delayed to 720 s for improved depiction of the lower ureter while opacification of other UUT segments are not sensitive to delay time. When low-dose furosemide is administered, excretory phase delay may be reduced to an average of 450 s.

The other CTU protocol is called the split-technique with considerably different protocols of contrast bolus. The main idea is in the administration of one bolus of contrast followed by a variable delays of 480-1,000 s (recent practices report 600-660 s delay) and then followed by the injection of a second contrast bolus. After a constant delay of 90-120 s from the second bolus, an abdominal scan is acquired and as the first injected contrast is already excreted, the acquisition contains combined nephrographic and excretory phases in one scan therefore reducing radiation dose. Further modifications of the split-bolus technique includes triple-bolus contrast injection for the acquisition of combined corticomedullary-nephrographic-excretory phase data some 510 s after start of the first bolus with or without low-dose diuretics‬‬‬‬‬‬‬‬ ‬‬‬‬‬‬‬‬‬‬ Imaging of the UUT with MRI is challenging and, as with other imaging modalities MRU, has its strengths and weaknesses. MRI is susceptible to various artefacts including chemical shift misregisteration, wraparound, phase-encoded motion and susceptibility artefacts, which might be more prominent at higher field strength‬. Furthermore standing wave and conductivity artifact ‬are noticed in obese or ascites patients at 3T imaging. Therefore good knowledge and experience of both normal anatomy and artefacts are a prerequisite for correct image interpretation. MRI is lengthy examination and needs patient cooperation. Breath-hold ultrafast sequences and the use of parallel imaging reduces imaging time and are useful to obtain high quality images and hence help reduce movement artifacts. It is also beneficial to raise the arms over the head during coronal imaging to prevent wraparound artifact. In the investigators' experience reader should be always familiar with the artefacts related to the enhanced excretion of urine such as void lines and turbulence artefacts especially in the dilated pelvis. The investigators also recommend imaging the UUT routinely in both axial and coronal planes during the excretory phase.‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬‬ The inability to visualize calcifications are considered as a limitation to the use of MRU in the evaluation of UUT stone disease. Indeed possible stone is visualized as a partial or complete intraluminal filling defect which is nonspecific and should be differentiated with blood clot or tumor. Nevertheless, a clot is usually hyperintense at unenhanced sequence and do not enhance after the administration of contrast and additionally the margins of the soft-tissue abnormality are usually irregular compared with the well-defined margins of calculi. Opposite to that a tumor will usually enhance. Therefore any MRU protocol should include both T2 and T1 sequences and the latter both pre- and postcontrast sequences. The failure to do so might result in misinterpretations, yet occasionally severe edema might be misinterpreted as of a possible tumo. Different results from the literature should be interpreted with caution because of the variability of used sequences and selection bias. Not all studies evaluating the performance of MRU use both T1 and T2 sequences and as previously mentioned, T2 sequences alone are insufficient to evaluate the cause of obstruction.

MRU was shown to be superior to IVU in the detection of UUT stones. MRU was found to be at least as accurate as helical CT in the evaluation of patients with acute flank pain. Also the presence of secondary signs of obstruction such as the perirenal edema on the side of symptoms are highly suggestive of acute obstruction and is better visualized at MRU than at CT. Yet CT gained wider acceptance: CT is widely available, accurate and rapid imaging modality in the evaluation of acute flank pain and stone disease. MRU is an acceptable substitute in cases where the use of radiation is not desired in special patient populations i.e. in children, young adults and pregnant patients.

Another limitation of MRU is in the slight underestimation of the size of ureteral stones compared to CT and IVU. Also, according to the published results, small ureteral stones can be occasionally missed in chronic obstructions, especially when the secondary signs of acute obstruction are absent to raise the suspicions of a stone disease. Additionally MRU is insensitive in the detection of small calyceal stones therefore cannot reliably evaluate the actual stone disease-burden of the calyceal system, yet small stones are rarely of clinical importance.

A comprehensive MRU protocol facilitates evaluation of the renal parenchyma, UUT, surrounding structures and if needed the renal vasculature. This "one-stop evaluation" approach is fully applicable with MRU which is additionally free from radiation. Additionally MR is superior to CT in that it provides better tissue contrast resolution and greater sensitivity for contrast enhancement. Therefore MRU became the secondary investigation of choice after US in pediatric UUT imaging. The European Society of Paediatric Radiology uroradiology task force and ESUR paediatric working group recommends to always consider MRU, when available, as a secondary investigation after US in applicable situations, with the main principle being to avoid CT whenever possible. The few accepted major indications for CTU in children being severe urinary tract trauma, complicated/equivocal urolithiasis (if high level US+KUB are not conclusive and if there is expected therapeutic impact).

The MRU protocol includes always Both T2 and T1 breath-hold sequences in coronal orientation as a minimum. Nevertheless there are no universally accepted consensus protocol. As a safe method the investigators believe that MRU protocols should not duplicate CTU protocols in comparison, but a comprehensive protocol with multiple acquisitions is most probably beneficial.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for CTU to rule out malignancy

Exclusion Criteria:

* GFR >45; BEnign conditions; Contrast allergy; Contraindications to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Percentage opacification score of different UUT segments using a comprehensive 3T MRU protocol in comparison with 3-phase CTU protocol. | through study completion, an average of 1 year
  The UUT will be devided into 6 regions: Upper calyces, lower calyces, pelvis, and upper, middle and lower ureter, and the percentage opacification of each segment will be scored visually using 6 percentage-categories. Results of the opacification scores will be compared between MRU and CTU.

SECONDARY OUTCOMES:
Performance of MRU in comparison to CTU | through study completion, an average of 1 year
  Pathological findings from CTU will be compared to MRU; i.e. for the presence of tumors, Stones, obstruction and its causes.

CONTACTS AND LOCATIONS:
Overall Officials: Ritva Vanninen, MD; PhD, Study Director — Kuopio University Hospital; University of Eastern Finland
Locations (1):
- Kuopio University Hospital, Department of Clinical Radiology, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared after manuscript submission

REFERENCES:
- [Derived] Sudah M, Masarwah A, Kainulainen S, Pitkanen M, Matikka H, Dabravolskaite V, Aaltomaa S, Vanninen R. Comprehensive MR Urography Protocol: Equally Good Diagnostic Performance and Enhanced Visibility of the Upper Urinary Tract Compared to Triple-Phase CT Urography. PLoS One. 2016 Jul 6;11(7):e0158673. doi: 10.1371/journal.pone.0158673. eCollection 2016. PMID 27384417